CLINICAL TRIAL: NCT07348666
Title: BRITE 2.0: A Just-in-time Adaptive Intervention for Suicide Safety Planning in Adolescents (ViraSafe RCT (SBIR Phase 2))
Brief Title: A Just-in-time Adaptive Intervention for Suicide Safety Planning in Adolescents
Acronym: ViraSafeRCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ksana Health (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Pittsburgh Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY25040094; R44MH135605 (NIH)
Record Dates: First submitted 2026-01-15; First posted 2026-01-16 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Suicide; Mental Health Disorder; Anhedonia
Keywords: depression; depressive disorder; mood disorder; mental disorders; suicidal behavior; suicidal thoughts; suicidal ideation
MeSH Terms: conditions — Suicide; Mental Disorders; Anhedonia; Depression; Depressive Disorder; Mood Disorders; Suicidal Ideation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The clinical assessor is masked to the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ViraSafe (Experimental): The new augmented app that combines BRITE coping skills and safety planning into the Vira behavior change platform
  Interventions: Behavioral: ViraSafe: Treatment pushes
- BRITE (Active Comparator): The original BRITE app that promotes self-monitoring and self-management by providing strategies to avoid or cope with triggers for suicidal urges and has been rigorously tested in clinical trials
  Interventions: Behavioral: BRITE

INTERVENTIONS:
Behavioral: ViraSafe: Treatment pushes — ViraSafe participants will complete a safety plan with their provider. Safety plan content will be editable and viewable throughout the intervention for both participants and their providers. Participants will be able to access the safety plan at any time in ViraSafe. Additionally, patients using ViraSafe will be prompted to complete a daily distress rating. ViraSafe uses automated algorithms (i.e., just in time adaptive intervention features) and user input from distress ratings to facilitate increased engagement with coping skills and pushes safety planning materials to users at periods of high risk (i.e., increases in emotional distress).
  In addition to the just-in-time reminders (i.e., nudges) pushed automatically by the system, through the Vira Pro platform, practitioners can schedule just-in-time reminders (i.e., "nudges") to arrive in the user's phone to support their behavior change plan.
  Arms: ViraSafe
Behavioral: BRITE — The BRITE app contains the teen's safety plan, links to videos of how to use coping strategies they indicated in their safety plan that have been useful for them (like guided mediation or deep breathing), a library of evidence-based and age-appropriate coping skills and strategies that the adolescent can learn more about, photos or videos that the adolescent has uploaded to the app, and includes a question asking them to rate their distress level in the moment: "What is your distress level right now?" (1 is "Least Distressed" to 5, which is "Most Distressed"). Then, the teen is asked to identify the feeling that fits their distress level via 12 emoji images: "Which feelings fit your distress level?" Based on adolescent's distress rate, the BRITE app suggests coping skills or "activities" for the adolescent to lower their distress level.
  Arms: BRITE

SUMMARY:
Despite efforts to prevent suicide, US rates are climbing, and suicide is the second leading cause of death amongst youth. Digital tools, especially personal smartphones, are promising avenues to address these issues and can be used to increase engagement with effective interventions such as suicide safety planning. The BRITE suicide safety planning app was developed on evidence-based principles and has undergone rigorous formative development and effectiveness evaluations. However, to optimize its functionality, commercial viability, and scale its implementation, issues related to user engagement needed to be addressed. This 3 month Pragmatic Randomized Trial will evaluate the impact of the ViraSafe app-an enhanced version of the BRITE suicide safety planning app-on improving engagement with coping skills and safety planning among suicidal adolescents by comparing its intervention components to those of the original BRITE app.

DETAILED DESCRIPTION:
ViraSafe is an augmented version of the BRITE app that integrates the BRITE coping skills and safety planning content into a module within the Vira behavior change platform. Vira, a digital behavior change platform developed by Ksana Health, consists of a smartphone app for patients, along with integrated web portals for practitioners and for healthcare administrators and supervisors. The platform collects self-report and passive data on smartphone usage patterns, such as language use, physical activity, sleep, social interactions, and screen time, and uses these insights to provide objective and continuous measurements of mental health indicators.

Upon downloading the Vira app and accessing the ViraSafe module, participants will complete a safety plan with their provider. Safety plan content will be editable and viewable throughout the intervention for both participants and their providers. Participants will be able to access the safety plan at any time in ViraSafe. Additionally, patients using ViraSafe will be prompted to complete a daily distress rating. ViraSafe uses automated algorithms (i.e., just in time adaptive intervention features) and user input from distress ratings to facilitate increased engagement with coping skills and pushes safety planning materials to users at periods of high risk (i.e., increases in emotional distress).

In addition to the just-in-time reminders (i.e., nudges) pushed automatically by the system, through the Vira Pro platform, practitioners can schedule just-in-time reminders (i.e., "nudges") to arrive in the user's phone to support their behavior change plan.

After undergoing study screening procedures and providing informed consent/assent, participants will complete the baseline assessment (60 minutes) which will occur virtually over video conference software or phone call.

Additional self-reports collected at patient visit will be requested through informed consent process as some overlap with what research team plans to administer. Self-reports will be retrieved for data analysis at the timepoints that align with the study timepoints. Self-reports will be administered by research staff if not available from a clinic's measurement-based care system.

Following Baseline assessments, participants will be randomized in a 1:1 allocation to receive ViraSafe or BRITE (50 in each arm). Randomization will be based on age, sex, and suicide symptoms. At a scheduled patient visit in their clinical settings, onboarding to assigned app will occur. Onboarding involves downloading their assigned app from Google Play Store or Apple App Store. Each app involves a trained clinician from their clinic setting collaboratively completing a safety plan. If a mental health clinician is not available for onboarding after Baseline, a research clinician will assist with onboarding.

At 1-month timepoint, participants will repeat the assessment interview (which will occur virtually over video conference software or phone call) and self-report measures with additional items assessing acceptability, usability, and satisfaction using the Technology Acceptance Model (TAM) and System Usability Scale (SUS) (total assessment duration: 60 minutes). At the 3-month timepoint, participants will repeat the assessment interview (which will occur virtually over video conference software or phone call) and self-report measures (total duration: 60 minutes).

20 adolescent participants or as many that are needed to reach saturation who received ViraSafe intervention arm will be selected to complete a qualitative exit interview to provide additional feedback on the intervention (60 minutes). The interview guide will be developed closer to the time of first exit interview and submitted for approval to the IRB prior to completing interviews.

ELIGIBILITY:
Inclusion Criteria:

Youth (minors):

* 13-17 years old
* Suicide attempt in the last year and ideation in the past month
* English fluency and literacy
* Parent or legal guardian willing and able to legally provide informed consent
* Receiving care at one of the study clinical settings with trained providers to onboard ViraSafe or BRITE safety plan

Youth (adults)

* 18-24 years old
* Recent suicide attempt or ideation with a plan
* English fluency and literacy
* Receiving care at one of the study clinical settings with trained providers to onboard ViraSafe or BRITE safety plan.

Exclusion Criteria:

Youth (minors):

* Unable to read/understand English
* Current manic or psychotic episode
* Development disability precluding comprehension of study procedures
* No routine access to a mobile phone, assessed by EHR review and during phone screen
* No eligible parent or legal guardian to provide informed consent

Youth (adults):

* Unable to read/understand English
* Current manic or psychotic episode
* Development disability precluding comprehension of study procedures
* No routine access to a mobile phone, assessed by EHR review and during phone screen

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proximal Engagement | 24 hours
  Engagement with the ViraSafe app (i.e., tapping on the push notification, patterns of accessing app features such as coping skills and safety plan) and BRITE app (daily dose rating, post rating after accessing coping skill, editing coping skill content)
Engagement with the apps | 3 months
  Engagement over the course of the trial will be measured through objective app usage metrics, including total number and frequency of features used.

SECONDARY OUTCOMES:
Technology Acceptance | 3 months
  Mixed methods feedback on acceptability, usability, and satisfaction, including the System Usability Scale and items adapted from the Technology Acceptance Model (TAM).
  System Usability Scale: 10 items -- Brooke, J(1996) Technology Acceptance Model: 12 Items - Adapted from Davis, (1989)
  Participants rate the extent to which they agree with each statement by circling a number from one to seven arranged horizontally beneath anchor point descriptions "Strongly Agree," "Neutral," and "Strongly Disagree.
Suicide Risk Factors: Columbia Suicide Severity Rating Scale (CSSRS) | 3 months
  Changes in suicide risk factors from baseline to 3 months assessed through the Columbia Suicide Severity Rating Scale (CSSRS).
  The C-SSRS is an assessment of suicidal thoughts and behaviors in clinical and research settings. The C-SSRS consists of 16 questions about suicidal thoughts and behaviors (the first 10 questions comprise the ideation subscale and the last 6 comprise the behavior subscale). This 5-item subscale ranges from a minimum of 0 (corresponding to no suicidal ideation) to a maximum of 5 (representing active suicidal ideation with plan and intent).
Suicidal Risk Factors: Reason for Living | 3 months
  The Reasons for Living (RFL) Inventory is a 48-item instrument that measures a range of beliefs potentially important as reasons for not committing suicide. The items are rated on 6-point Likert type scales based on how important each reason would be for living if suicide was contemplated (1 = not at all important; 6 = extremely important). The total score is calculating by calculating the mean of the item scores and multiplying the result by 48. Total scores can only be calculated if a participant answers at least 38 items.

OTHER OUTCOMES:
Depressive Symptoms: Mood and Feelings Questionnaire (MFQ) | 3 months
  Changes in self-reported depressive symptoms from baseline to 3 months, assessed through the Mood and Feelings Questionnaire (MFQ).
  The MFQ is a 13-item self-report questionnaire used to screen for depressive in children and young people. Items are rated on a 3-point Likert scale (not true = 0; sometimes true = 1; not true = 2). Scores are calculated by summing the point values on each response. Total MFQ scores range from 0 to 26, with higher scores suggesting greater severity in depressive symptoms.
Anxiety Symptoms: the Screen for Anxiety Related Emotional Disorders (SCARED) | 3 months
  Changes in self-reported anxiety symptoms from baseline to 3 months, assessed through the Screen for Anxiety Related Emotional Disorders (SCARED)
  The SCARED is a 5-item self-report questionnaire used to screen for childhood anxiety disorders including general anxiety disorder, separate anxiety disorder, panic disorder, and social phobia. Items are rated on a 3-point Likert scale from 0 to 2 and summed to yield a total score. Total scores range from 0 to 10. Higher scores indicate greater anxiety.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Ksana Health Inc, Eugene, Oregon
  - STAR Center, Western Psychiatric Institute & Clinic, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania